CLINICAL TRIAL: NCT00610259
Title: Brief Behavioral Therapy for Insomnia (bBT-I) for Depressed Outpatients With Refractory Insomnia - An Assessors-blinded, Randomized Controlled Effectiveness Trial
Brief Title: Brief Behavioral Therapy for Insomnia (bBT-I) for Depressed Outpatients With Refractory Insomnia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nagoya City University (Other)
Collaborators: Kochi University (Other)
Responsible Party: Toshiaki Furukawa, Nagoya City University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCUPsychiatry001; HLSRG (Ministry of Health)
Record Dates: First submitted 2008-01-16; First posted 2008-02-07 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Major Depressive Disorder
Keywords: Depressive disorder; Sleep initiation and maintenance disorder; Behavior therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): brief behavioral therapy for insomnia (bBT-I) in addition to treatment as usual (TAU)
  Interventions: Behavioral: brief behavioral therapy for insomnia (bBT-I); Other: Treatment as usual (TAU)
- 2 (Active Comparator): Treatment as usual (TAU)
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: brief behavioral therapy for insomnia (bBT-I) — 4 50-minute individual sessions every week for 4 weeks
  Arms: 1
Other: Treatment as usual (TAU) — The psychiatrist-in-charge sees the patient once every 2 weeks for approximately 10 minutes each to monitor pharmacotherapy.

SUMMARY:
The purpose of this study is to examine the effectiveness of brief behavioral therapy for insomnia (bBT-I) in addition to treatment as usual (TAU) in comparison with TAU alone for refractory insomnia among patients with major depression in partial remission.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV major depressive disorder, as ascertained by the Structured Clinical Interview for DSM-IV Axis I disorders (SCID)
2. Either sex, between 20 and 70 years of age at the time of entry into the trial
3. Outpatient at the time of entry into the trial
4. For the index episode, patients have to have already been on two types of adequate doses of antidepressants for no shorter than 4 weeks for each medication or already on two types of antidepressants for 8 weeks in total even if the doses of the drugs have not been adequate due to side effects. The medication has not been changed for at least 4 weeks prior to the study entry.
5. A score of 2 on at least one of the three sleep items of the 17-GRID-HAMD and a score of 8 or more on the ISI.
6. A score between 8 and 23 on the 17-GRID-HAMD.
7. Agreement to the requirements that i) no change of medication will be allowed during the first 4 weeks of their study period, and ii) all the treatment sessions both of bBT-I and of TAU will be audiotaped for the purpose of checking their adherence to the protocol

Exclusion Criteria:

1. Their mental or physical status at the time of entry into the trial is regarded as so critical as to need immediate hospitalisation
2. A serious suicidal risk, defined as a score of 3 or more on item 3 (suicidal ideation) of the 17-GRID-HAMD
3. Patients who have had or are having any structured psychotherapy (e.g. cognitive therapy, or family therapy) at the time of entry
4. Patients with current diagnosis of primary anxiety or personality disorder, insomnia associated with another sleep disorder, significant medical problems, current drug or alcohol substance abuse or dependence, or psychosis, or with a history of schizophrenia or bipolar disorder
5. Patients with duration of depression shorter than 2 months
6. Their insomnia is considered to derive from sleep apnoea or periodic limb movements during sleep, judged by their clinicians.
7. Patients who engage in work involving night-shift, which might influence sleep status
8. Patients currently taking methylphenidate or modafinil.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Changes in the total Insomnia Severity Index (ISI) score between the baseline and the 8-week assessment | at 8-week

SECONDARY OUTCOMES:
"No clinically significant insomnia" at the 8-week assessment, which is defined as 7 or less on the total ISI score | at 8-week
"No clinically significant insomnia" at the 4-week assessment, which is defined as 7 or less on the total ISI score | at 4-week
Changes in the total ISI score between the baseline and the 4-week assessment | at 4-week
Changes in the total score of the modified Pittsburgh Sleep Quality Index (PSQI) between the baseline and the 8-week assessment | at 8-week
Changes in the total score of the modified PSQI between the baseline and the 4-week assessment | at 4-week
Changes in the 17-item Hamilton Rating Scale for Depression (HAMD) between the baseline and the 8-week assessment | at 8-week
Changes in the 17- HAMD between the baseline and the 4-week assessment | at 4-week
Changes in the Short Form 36 (SF-36) scores between the baseline and the 8-week assessment | at 8-week
Changes in the SF-36 scores between the baseline and the 4-week assessment | at 4-week

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki A Furukawa, MD, PhD, Principal Investigator — Nagoya City University Graduate School of Medical Sciences
Locations (1):
- Nagoya City University Graduate School of Medical Sciences, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Derived] Shimodera S, Watanabe N, Furukawa TA, Katsuki F, Fujita H, Sasaki M, Perlis ML. Change in quality of life after brief behavioral therapy for insomnia in concurrent depression: analysis of the effects of a randomized controlled trial. J Clin Sleep Med. 2014 Apr 15;10(4):433-9. doi: 10.5664/jcsm.3624. PMID 24733990
- [Derived] Watanabe N, Furukawa TA, Shimodera S, Morokuma I, Katsuki F, Fujita H, Sasaki M, Kawamura C, Perlis ML. Brief behavioral therapy for refractory insomnia in residual depression: an assessor-blind, randomized controlled trial. J Clin Psychiatry. 2011 Dec;72(12):1651-8. doi: 10.4088/JCP.10m06130gry. Epub 2011 Mar 8. PMID 21457679